CLINICAL TRIAL: NCT06277544
Title: Analysis of Prognosis and Risk Factors of Lateral Ankle Ligament Reconstruction Procedure for Patients With Avulsion Fracture of the Lateral Ankle Ligament: a Prospective Cohort Study
Brief Title: Analysis of Prognosis and Risk Factors of LAL Reconstruction Procedure for Patients With AF of the LAL: a Prospective Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2024087
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-01

CONDITIONS: Avulsion Fracture of Lateral Ankle Ligament
MeSH Terms: interventions — Plastic Surgery Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- rupture group: rupture of lateral ankle ligament
  Interventions: Procedure: lateral ankle ligament repair or reconstruction
- fracture group: avulsion fracture of lateral ankle ligament
  Interventions: Procedure: lateral ankle ligament repair or reconstruction

INTERVENTIONS:
Procedure: lateral ankle ligament repair or reconstruction — repair or reconstruction procedure for lateral ankle ligament

SUMMARY:
To compare the clinical outcomes of CAI patients with and without lateral ankle avulsion fracture after ligament repair/reconstruction, and to analyze the risk factors associated with the outcome.

DETAILED DESCRIPTION:
80 patients with external ankle ligament injury without avulsion fracture and 40 patients with external ankle ligament injury combined with avulsion fracture were treated by surgery in our department. The outcomes included Karlsson score, VAS, AOFAS and Tegner score. The outcomes were compared between the two groups, and the risk factors were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years old
2. Chronic pain or instability in the ankle, injury to the lateral collateral ligament of the ankle determined by MRI examination of the ankle, and distal avulsion fracture of the fibula indicated by CT examination.
3. Patients with poor results after more than 3 months of conservative treatment with rest/topical/oral non-steroidal anti-inflammatory drugs
4. Patients voluntarily participate in clinical trials, sign informed consent, and can cooperate with clinical follow-up

Exclusion Criteria:

1. Persons who have participated in clinical trials of other drugs or medical devices within the last 6 months
2. Malalignment of ankle joint force (varus or valgus >5 degrees)
3. Chronic specific synovitis (rheumatoid, pigmented villonodular synovitis, etc.)
4. Patients with joint fibrosis, joint stiffness, and obvious limited movemente. Moderate to severe osteoarthritis (Takakura stage III or IV)

f. Patients with contraindications to MRI g. Hemophiliacs h. Patients with systemic conditions that cannot tolerate surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with chronic lateral ankle instability with or without lateral ankle avulsion fracture meeting surgical indications.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-01-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Karlsson score | 2 weeks, 3 months, 6 months, 1 year, and 2 years
  The Karlsson score consists of seven questions covering ankle pain, swelling, levels of daily activity and exercise .et al,provided by the patient with objective scores. The minimum and maximum values of Karlsson are 0 and 100, respectively. And higher scores mean a better outcome

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | 2 weeks, 3 months, 6 months, 1 year, and 2 years
  The Visual Analogue Scale (VAS) is designed to present to the respondent a rating scale with minimum constraints. Respondents mark the location on the 10-centimeter line corresponding to the amount of pain they experienced. This gives them the greatest freedom to choose their pain's exact intensity. It also gives the maximum opportunity for each respondent to express a personal response style. The minimum and maximum values of VAS are 10 and 0, respectively. And higher scores mean a worse outcome.
American Orthopaedic Foot and Ankle Society (AOFAS) | 2 weeks, 3 months, 6 months, 1 year, and 2 years
  The American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Score combines subjective scores of pain and function provided by the patient with objective scores based on the surgeon's physical examination of the patient (to assess sagittal motion, hindfoot motion, ankle-hindfoot stability and alignment of the ankle-hindfoot). The scale includes nine items that can be divided into three subscales (pain, function and alignment). The minimum and maximum values of AOFAS are 100 and 0, respectively. And higher scores mean a better outcome.
Tegner Scale | 2 weeks, 3 months, 6 months, 1 year, and 2 years
  The Tegner Scale is a tool commonly used to assess the degree of sports injury and the degree of functional recovery, which is graded according to the level of motor activity a participant participates in and the gradual increase in requirements. It is graded on a scale of 0 to 10, with the specific meanings.

CONTACTS AND LOCATIONS:
Overall Officials: Guo Qinwei, MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided